CLINICAL TRIAL: NCT01835535
Title: Clinical Evaluation of the Therapeutic Intra-Vascular Ultrasound (TIVUS™) System for Renal Denervation in Patients With Resistant Hypertension
Brief Title: Continued Safety and Performance of the TIVUS System
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cardiosonic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN02-001
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Hypertension, Resistant to Conventional Therapy
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Severe Resistant HTN (Experimental): Patients presenting with resistant hypertension and office systolic blood pressure of 160 mmHg (150 mmHg for DM) or greater
  Interventions: Device: TIVUS

INTERVENTIONS:
Device: TIVUS

SUMMARY:
The TIVUS II is a prospective, multicenter, non-randomized, open-label clinical study of the safety and performance of the TIVUS™ System consisting of three (3) concurrent cohorts:

* TIVUS™ Severe Resistant HTN Cohort
* TIVUS™ Moderate Resistant HTN Cohort
* TIVUS™ Failed RF Therapy Cohort

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 and ≤ 80 years of age
* For Cohort A: Documented office systolic blood pressure > 160 mmHg (> 150 mmHg for diabetic patients); For Cohort B: Documented office systolic blood pressure > 140 mmHg (> 130 mmHg for diabetic patients); For Cohort C: Documented office systolic blood pressure > 150 mmHg (> 140 mmHg for diabetic patients)
* Documented 24 hour systolic ABPM > 135 mmHg
* Adherence to a stable drug regimen
* For patients in Cohort C only: Documented renal denervation procedure with any RF technology 12 months or more prior to screening
* Suitable renal artery anatomy
* Male or non-pregnant / non-lactating female
* Patient understands the nature of the procedure and provides written informed consent
* Patient is willing and able to comply with the specified study requirements and follow-up evaluations

Exclusion Criteria:

* eGFR < 45mL/min/1.73m2
* Documented primary pulmonary hypertension
* Patient experienced >1 episode of orthostatic hypotension coupled with syncope
* Documented indicator of a secondary renal hypertension
* History of myocardial infarction, unstable angina pectoris, or a cerebrovascular accident within 6 months
* Planned major surgery or cardiovascular intervention in the next 6 months
* Surgery or cardiovascular intervention in the previous 3 months
* Hemodynamically significant valvular heart disease
* Severe debilitating lung disease
* Patient on anticoagulant therapy that cannot be temporarily withheld for performing catheterization
* Patient has a single functioning kidney
* Documented thrombocytopenia, clotting disorders or aortic aneurysms
* Moribund patient, or patient with comorbidities limiting life expectancy to less than one year
* Contraindication to recommended study medications or intravascular contrast material that cannot be adequately controlled with pre-medication
* Concurrent enrollment in another trial
* Main renal arteries < 4 mm in lumen diameter or < 20 mm in length
* Aorto-renal angle that prevents a safe cannulation of the renal artery
* Severe common femoral artery, common and/or external iliac artery, renal, iliac or aortic calcification or tortuosity that may compromise the safe performance and completion of the procedure
* Hemodynamically or anatomically significant renal artery abnormality or stenosis in either renal artery
* Any renal artery stenosis > 50% by visual assessment
* Any renal artery aneurysm in either renal artery
* A history of prior renal artery balloon angioplasty or stenting (for patients in Cohort A and B only, also a history of prior renal denervation at any time)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in office Systolic Blood Pressure (SBP) from baseline to 6-month | 6 month

SECONDARY OUTCOMES:
Procedural complications | 30 day
Major Adverse Events (MAE) | 1 year
Preservation of renal function | 1 year
Cardiovascular complications | 1 year
Blood pressure reduction | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jonas, MD, Principal Investigator — Kaplan Medical Center
Locations (1):
- Royal Perth Hospital, Perth, Australia